CLINICAL TRIAL: NCT05444348
Title: Compassionate Communication and Advance Care Planning to Improve End of Life Care in Treatment of Hematological Disease (ACT)- a Cluster Randomized Controlled Study
Brief Title: Compassionate Communication and Advance Care Planning to Improve End of Life Care in Treatment of Hematological Disease (ACT)
Acronym: ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christoffer Johansen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Vejle Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Gødstrup Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Christoffer Johansen, Professor MD, PhD, DMsc (Med), Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2022-93
Record Dates: First submitted 2022-05-19; First posted 2022-07-05 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma; Acute Myeloid Leukemia
MeSH Terms: conditions — Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma; Leukemia, Myeloid, Acute | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT intervention (Experimental): Participants will receive the ACT intervention
  Interventions: Behavioral: Advance consultation concerning your life and treatment (ACT )
- control (No Intervention): Participants will receive no intervention only usual care.

INTERVENTIONS:
Behavioral: Advance consultation concerning your life and treatment (ACT ) — The ACT intervention consists of: an 8 h training day for clinicians including clinical materials such as a conversation aid and conversations guide. 6o minutes ACT-intervention sessions in daily clinic. the patients and caregivers will receive preparatory material prior for the ACT-intervention sessions, and a 30 min follow-up telephone call from the nurse within one week after the ACT-session. Clinicians will receive five sessions of followup supervision within the 24 months of intervention. The 60 min ACT-intervention session is an interdisciplinary conversation with nurse, physician, patient, and caregiver discussing issues of importance of patient and caregiver. The issues are based on the preparatory material focusing on information level and prognosis, patient's and caregiver's values, hopes, fears and worries regarding the future care with progressive disease.
  Arms: ACT intervention

SUMMARY:
Patients diagnosed with hematologic cancer are at substantial risk of dying, as 5-year survival among patients with acute myeloid leukemia is 20 % and only every second patient treated for incurable myeloma lives 5 years after date of diagnosis. Nevertheless, many overestimate their prognosis, and value of therapy. Patients with hematological cancers frequently have poor end of life outcomes, such as high treatment activity close to death, where clinical effects are doubtful, and low utilization of palliative care. Prognostic awareness and end of life (EOL) issues have urgency in the communication between patients, their caregiving relatives, and clinicians, in order to avoid futile treatments and suffering at EOL. Inspired by advanced care planning, the investigators developed the concept "Advance Consultations Concerning participants Life and Treatment" (ACT) in collaboration with a group consisting of hematologists, nurses, patients, and caregivers. The ACT concept consists of an 8-hour training day for clinicians, clinical tools, system changes, and preparation material for patients and caregivers prior to the consultation. ACT involves patients and caregivers earlier in preparation for life with chronic progressive disease and EOL-decisions, through an intervention based on compassionate communication and early planning of EOL-care. The aim of the study is to investigate the effect of the intervention on use of chemotherapy and quality of EOL-care in patients with hematological malignancy. Based on the results of the completed pilot study, the investigators are planning a nationwide 2-arm cluster randomized controlled trial where 40 physicians and 80 nurses across seven different hematological departments are randomized to either usual care or ACT training and completing ACT conversations. The investigators expect to include a total of 400 patients and their family caregivers. It is hypothesized that the ACT intervention will decrease use of futile chemotherapy, prepare patients and caregivers for difficult end-of-life-decisions, and improve quality of end-of-life care in hematology.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

* Be at least 18 years of age
* Have a diagnosis of one of the following:
* High-risk myelodysplastic syndrome (MDS) or MDS with overlap of myeloproliferative neoplasms (high-risk MDS/MPN),
* Acute myeloid leukemia(AML): Age≥80 or in palliative treatment or relapse
* Lymphoma: Age≥80 or relapse or refractory or palliative treatment
* Multiple myeloma(MM): Age≥80 or relapsed or refractory

Have limited treatment options. Provide informed consent. Have sufficient Danish skills to complete intervention sessions and data collection

An informal caregiver is identified by the patient as the primary provider of informal physical, practical or emotional support and must:

* Be at least 18 years of age
* Be able to accompany patients to intervention appointments
* Provide informed consent
* Have sufficient Danish skills to complete intervention sessions and data collection

Physicians:

* specialized in hematology
* treating patients with High risk myelodysplastic syndrome, acute myeloid leukemia, lymphoma, or multiple myeloma
* work at the same department for the entire time of intervention.

Nurses:

* treating patients with High-risk myelodysplastic syndrome, acute myeloid leukemia, lymphoma, or multiple myeloma
* work at the same department for the entire time of intervention.

Exclusion Criteria:

Patient and caregiver are excluded if one of them is:

- Suffering from a severe psychiatric disorder

Physicians and nurses:

- If they do not meet the inclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Use of chemotherapy within the last 30 days of life. | 30 days prior to date of death, if patient dies within 18 months of follow-up period of the study
  Counts of patients receiving chemotherapy in the last 30 days of their life
Change from baseline through 3,6,9,12 and 18 months follow-up in patient's anxiety symptoms | baseline, 3,6,9,12, and 18 months of follow-up. Investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Patient reported outcome of anxiety (General anxiety disorder), reporting on a 4-point scale from 0-3 with high value as worse outcome.
Change from baseline through 3,6,9,12 and 18 months follow-up in caregiver's anxiety symptoms | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Caregiver reported outcome of anxiety (General anxiety disorder), reporting on a 4-point scale from 0-3 with high value as worse outcome.

SECONDARY OUTCOMES:
Number of Days of hospitalized in the last 30 days of life | 30 days prior to date of death, if patient dies within 18 months of follow-up period of the study
  Counts of days in hospital in the last 30 days of life of deceased patients
Number of medical consultations, in the last 30 days of life | 30 days prior to date of death,if patient dies within 18 months of follow-up period of the study
  Counts of medical consultation in the last 30 days of life of deceased patients
Number of patients with referral to hospice in the last 30 days of life | 30 days prior to date of death, if patient dies within 18 months of follow-up period of the study
  Referral to hospice and days from referral to death
Survival | days from diagnosis to death, if patient dies within 18 months follow-up period of the study
  Overall survival
Change from baseline through 3,6,9,12 and 18 months follow-up in Patient's quality of life | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Patient reported outcome using European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire Core 15 item palliative, 4-point scale, minimum value: 1 max value 4, higher score worse outcome
Change from baseline through 3,6,9,12 and 18 months follow-up in patients' depressive symptoms | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Patient reported outcome of depression (patient Health Questionaires), reporting on a 4-point scale from 0-3 with high value as worse outcome.
Change from baseline through 3,6,9,12 and 18 months follow-up in caregivers' depressive symptoms | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Caregiver reported outcome of depression (patient Health Questionaires), reporting on a 4-point scale from 0-3 with high value as worse outcome.
Change from baseline through 3,6,9,12 and 18 months follow-up in patient's social support | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated mea
  Patient reported outcome, questionnaire: Ways of providing support, 19-item, measure on a 5-point scale ranging from "never" to "very often"
Change from baseline through 3,6,9,12 and 18 months follow-up in caregiver's social support | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated mea
  Caregiver reported outcome, questionnaire: Ways of providing support, 19-item, measure on a 5-point scale ranging from "never" to "very often"
Change from baseline through 3,6,9,12 and 18 months follow-up in patient's relationship quality | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated mea
  Patient reported outcome, questionnaire: Relationship ladder, single-item, measure on a scale from 0-10, with higher value as better quality
Change from baseline through 3,6,9,12 and 18 months follow-up in caregiver's relationship quality | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated mea
  Caregiver reported outcome, questionnaire: Relationship ladder, single-item, measure on a scale from 0-10, with higher value as better quality
Change from baseline through 3,6,9,12 and 18 months follow-up in patient's satisfaction with health care | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Patient reported outcome: Family Satisfaction With Advanced Cancer Care, measure on a 5-point scale where 1 is best and 5 is worst.
Change from baseline through 3,6,9,12 and 18 months follow-up in caregiver's satisfaction with health care | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Caregiver reported outcome: Family Satisfaction With Advanced Cancer Care, measure on a 5-point scale where 1 is best and 5 is worst.
Change from baseline through 3,6,9,12 and 18 months follow-up in patient's prognostic understanding | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Patient reported outcome: Prognostic understanding, single item questionnaire
Change from baseline through 3,6,9,12 and 18 months follow-up in caregiver Prognostic understanding | baseline, 3,6,9,12, and 18 months of follow-up. investigator will use mixed effects models to utilize the repeated measurements at 3, 6, 9, 12, and 18, months follow-up.
  Caregiver reported outcome: Prognostic understanding, single item questionnaire
Patient satisfaction with intervention sessions | 7 days after each ACT intervention session through the study until 8 months of follow-up for intervention group
  Patient reported outcome: Satisfaction with intervention sessions, questionnaire developed for the intervention, 5 point scale from 1-5, higher score is better outcome.
Caregiver Satisfaction with intervention sessions | 7 days after each ACT intervention session through the study until 8 months of follow-up for intervention group
  Caregiver reported outcome: Satisfaction with intervention sessions, questionnaire developed for the intervention, 5 point scale from 1-5, higher score is better outcome.
Bereaved caregivers' depressive symptoms | 1 and 6 months after patient's death, if the patient dies within 18 months follow-up period of the study.
  Caregiver reported outcome of depression (patient Health Questionaires), reporting on a 4-point scale from 0-3 with high value as worse outcome.
Bereaved caregivers' anxiety symptoms | 1 and 6 months after patient's death, if the patient dies within 18 months follow-up period of the study
  Caregiver reported outcome of anxiety (General anxiety disorder), reporting on a 4-point scale from 0-3 with high value as worse outcome.
Post-traumatic stress | 1 and 6 months after patient's death, if patient dies within 18 months of follow-up period of the study
  Bereaved caregiver reported outcome: post-traumatic stress using questionnaire "Impact of Events Scale- revised", assesses subjective distress caused by traumatic events, Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Higher score worse outcome
Perception of the patient's quality of death | One months after patient's death, if patient dies within 18 months of follow-up period of the study
  Bereaved caregiver reported outcome: Perception of the patient's quality of death, The Views Of Informal Carers - Evaluation of Services - Short Form.
Prolonged Grief | six months after patient's death, if patient dies within 18 months of follow-up period of the study
  Bereaved caregiver reported outcome: Prolonged Grief disorder. using a 5-point scale from 1-5, Higher score means worse outcome
Self-efficacy - advance care planning | Baseline, and after completion of 5 ACT-intervention sessions (intervention group) through study completion, an average of 1 year, and after 24 months of intervention.
  Clinician reported outcome: Advance care planning self-efficacy, 5 point scale from 1-5, higher score is better outcome
Burnout | Baseline, and after completion of 5 ACT-intervention sessions (intervention group) through study completion, an average of 1 year, and after 24 months of intervention.
  Clinician reported outcome: burnout (Copenhagen Burnout Inventory) 5-point scale, value 0-5, higher score means worse outcome
Existential communication | Baseline, and after completion of 5 ACT-intervention sessions (intervention group) through study completion, an average of 1 year, and after 24 months of intervention.
  Clinician reported outcome: Existential communication, 5 point scale from 1-5, higher score is better outcome.
Satisfaction with intervention | After completion of 5 ACT-intervention sessions (intervention group) through study completion, an average of 1 year,
  Clinician reported outcome: satisfaction with intervention, questionnaire developed for the intervention, 5 point scale from 1-5, higher score is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (7):
- Denmark (7):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Sydvestjysk sygehus - Esbjerg, Esbjerg
  - Regionshospitalet Gødstrup, Herning
  - Odense Universitetshospital, Odense
  - Sjællands universitetshospital Roskilde, Roskilde
  - Lillebælt syge - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Access to protocol and statistical code, as well as Individual participation data (IPD) for meta-analysis will be possible upon request. Data requestors will need to sign a data access agreement in agreement with the Data Protection Act.
Supporting Information: Study Protocol, Analytic Code

REFERENCES:
- [Derived] Borregaard Myrhoj C, Clemmensen SN, Jarden M, Johansen C, von Heymann A. Compassionate Communication and Advance Care Planning to improve End-of-life Care in Treatment of Haematological Disease 'ACT': Study Protocol for a Cluster-randomized trial. BMJ Open. 2024 May 21;14(5):e085163. doi: 10.1136/bmjopen-2024-085163. PMID 38772898